CLINICAL TRIAL: NCT05028608
Title: Open-label, Fixed Sequence Crossover Study to Investigate the Effects of Carbamazepine on the Pharmacokinetics of Elinzanetant (BAY 3427080) in Healthy Participants.
Brief Title: A Study to Learn What Happens to Elinzanetant in the Body When Taken With or Without Carbamazepine, and How Safe it is in Healthy Men and Women Aged 18 to 60 Years.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21667; 2021-000309-26 (EudraCT Number)
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Vasomotor Symptoms as a Sex Hormone-dependent Disorder in Women and Men
Keywords: Vasomotor symptoms,; Menopause,; Healthy volunteers.
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Midazolam; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): Fixed treatment sequence starting with 2 single oral doses of midazolam and a single dose of elinzanetant.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Midazolam
- Period 2 (Experimental): Up titration of carbamazepine over 4 days (dose 1, 2, 3) continued by fixed dose 3 of carbamazepine prior to administration of midazolam / elinzanetant, followed by carbamazepine administration.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Midazolam; Drug: Carbamazepine

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — Elinzanetant given orally as a single dose in Period 1 and in Period 2.
  Other Names: NT-814
Drug: Midazolam — Midazolam given orally as single dose in Period 1 and in Period 2.
Drug: Carbamazepine — Carbamazepine given orally twice daily in Period 2 .
  Arms: Period 2

SUMMARY:
Researchers are looking for a better way to treat people who have symptoms caused by hormonal changes, such as hot flashes. Before a treatment can be approved for patients to take, researchers do clinical studies to better understand its safety and what happens to the treatment in the body.

In this study researchers want to learn more about a new substance called elinzanetant.

Elinzanetant, the study treatment, was developed to treat symptoms caused by hormonal changes, such as hot flashes. Carbamazepine is a drug that is already available for doctors to prescribe, for example against seizures. Midazolam is a treatment that is already available for doctors to prescribe as a sedative (calming treatment) or to help people sleep.

In this study, the researchers will learn how much elinzanetant gets into the participants' blood when taken with or without carbamazepine. They will also get to know if taking elinzanetant will affect the amount of midazolam in the blood.

The participants will all take elinzanetant as capsules, carbamazepine as tablets and midazolam as a liquid by mouth. On some days, they will take only 1 treatment of midazolam or carbamazepine or only elinzanetant. On other days, they will take two study treatments. On 3 different days during the study, the participants will take elinzanetant with midazolam, elinzanetant with carbamazepine and midazolam with carbamazepine.

Each participant will be in the study for up to 10 weeks. But, the entire study will last about 4 months.

During the study, all of the participants will stay at the study site for 2 periods, period 1 with 9 overnight stays and period 2 with 22 overnight stays at the study site. In addition, there will be two ambulatory visits, one before joining the study and one at the end of the study.

Blood and urine samples will be collected. The doctors will also check the participants' heart health using an electrocardiogram (ECG). The participants will answer questions about how they are feeling and about any medications they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 60 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG), vital signs, respiratory rate and body temperature.
* Body weight above or equal 50 kg and body mass index (BMI) within the range 18.0 and 30.0 kg/m^2(inclusive).
* Male and female:

Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

* Male participants: Male participants of reproductive potential must agree to use a condom (with or without spermicide) when sexually active. This applies for the time period between the signing of the informed consent form (ICF) until 5 days after the last dose of study intervention. Female partners of childbearing potential of male participants do not need to follow special precautions.
* Female participants: Women of childbearing potential will have to use highly effective non-hormonal contraception when having sexual intercourse with a male partner from signing the ICF until 5 days after last dose of the study drug. Women of non-childbearing potential are not required to use contraception.

Exclusion criteria

* Any clinically relevant abnormal findings in medical history and physical examination which in the opinion of the investigators, may put the participant at risk because of his/her participation in the trial or provide difficulties in interpreting the trial data.
* Known hypersensitivity to the study interventions (active substances, or excipients of the preparations), or structurally related drugs to CBZ (carbamazepine, e.g. tricyclic antidepressants).
* History of bone marrow depression.
* History of clinically hepatic disorders including hepatic porphyria (e.g. acute intermittent porphyria, variegate porphyria, porphyria cutanea tarda).
* History or family history of severe cutaneous reactions including toxic epidermal necrolysis and Stevens-Johnson syndrome.
* Human leukocyte antigen A (HLA-A) *31:01 or human leukocyte antigen B (HLA-B) *15:02 allele.
* History of myotonic dystrophy.
* History of clinically relevant psychiatric disorder, including psychosis or latent psychosis.
* History of epileptic seizures.
* History of clinically relevant depression, or suicidal ideation or behavior.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
AUC of elinzanetant with carbamazepine. | Period 2: Predose, Day 1 to Day 8
  AUC: Area under the concentration vs. time curve from zero to infinity after single (first) dose.
AUC of elinzanetant without carbamazepine. | Period 1: Predose, Day 1 to Day 8
  AUC: Area under the concentration vs. time curve from zero to infinity after single (first) dose.
Cmax of elinzanetant with carbamazepine. | Period 2: Predose, Day 1 to Day 8
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration.
Cmax of elinzanetant without carbamazepine. | Period 1: Predose, Day 1 to Day 8
  Cmax: Maximum observed drug concentration in measured matrix after single dose administration.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) without concomitant carbamazepine. | After the first administration of study intervention up to 7 days after the last administration
Number of participants with TEAEs with concomitant carbamazepine. | After the first administration of study intervention up to 7 days after the last administration

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data later will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.